CLINICAL TRIAL: NCT03606265
Title: The Effectiveness of a Web-based App for the Treatment of Chronic Pain
Brief Title: Utility of a Web-based App for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: HOSPITAL GENERAL UNIVERSITARIO DE CASTELLÓ (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GeneralAPP
Record Dates: First submitted 2018-06-27; First posted 2018-07-30 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App+Web (Experimental): Treatment as usual + app Participants at this condition will receive the usual medical treatment for their pain but also they will be monitored daily using the Pain Monitor app. Alarms will be generated in the face of certain preestablished events. Physicians will be asked to call patients and change/stop treatment if an alarm is received.
  Interventions: Device: App+Web
- Treatment as usual (Active Comparator): Treatment as usual (waiting list) Patients at this condition will receive the usual medical treatment at the pain unit, but they will not be monitored daily using the app.
  Interventions: Device: Treatment as usual

INTERVENTIONS:
Device: App+Web — Patients will use an app daily twice and physicians will use a website to consult the characteristics of the alarms the app will send them in the presence of an unwanted event
  Arms: App+Web
Device: Treatment as usual — Patients will be offered the usual treatment for their pain, which is not changed by study participation
  Arms: Treatment as usual

SUMMARY:
This study will compare the effectiveness of a web-based app compared to the treatment as usual without an app for the telemonitoring of patients with chronic pain. Two conditions will be set:

1. usual treatment (waiting list)
2. usual treatment + app

DETAILED DESCRIPTION:
Chronic pain is defined as one that lasts for at least three to six months, provided that this time is greater than the normal healing period of an injury. This pathology has become an important public health problem due to its high prevalence. In particular, it is estimated that it affects 20-30% of the adult population around the world. Medical interventions are the first-line treatment in recent clinical practice guidelines. Unfortunately, the effectiveness of medical interventions is only modest. Treatments significantly reduce pain on average, but the effect tends to be small . In addition, the drugs are not effective for a large percentage of patients. What these and other research suggest is that focusing only on large sample studies and the use of average change scores calls into question the usefulness of current patient-centered treatments. As noted by Dr. Turk, when data are averaged, various pain syndromes, drugs, surgical procedures, and studies in different countries are often included, which may mask the efficacy results of different treatments with Different samples. Single case methodology could be one of the ways to overcome these limitations. The single case investigation is a type of experimental study that offers experimental control within a single case. Some studies have already demonstrated the usefulness of these designs in chronic pain. In fact, the benefits of using this methodology as opposed to large sample studies were discussed recently during the 10th Congress of the European Pain Federation. These benefits include the need for a reduced number of participants, the ability to follow clinical evolution in real time and continuously, the amount of data provided, and applicability when using a control group is impractical or unethical. The investigators conducting the present investigation recently conducted a study at the Pain Unit of the Hospital General de Castellón to explore the effectiveness of current medical treatments. According to previous investigations, the treatment effect was only small (d = 0.32) and only a percentage of the patients (18.1%) had a clinically significant reduction of pain (ie a reduction greater than 30% ). From these results and the literature reviewed, a single case design could be an alternative method for research in the Pain Unit. However, the implementation of this type of methodology can be very costly due to the continuous evaluation of the evolution of the patient. In this sense, several studies have already shown that mobile applications (app) can effectively control the evolution of a wide range of pathologies in health settings . In fact, a recent controlled clinical study found that ecological records performed with mobile app had greater reliability than paper-and-pencil records. Rosser and Eccleston conducted a comprehensive review of existing apps for pain and the conclusion was that there was little evidence to support the use of current apps. Specifically, these authors showed that most apps did not specify whether their content was validated, did not include psychological components and none had been applied in a clinical study. In light of these results, Dr. Carlos Suso Ribera and Dr. Ribera Canudas contacted the research team Labpsitec of Jaume I University, who were developing an application for pain called "Pain Monitor". Dr. Carlos Suso Ribera and Dr. Ribera Canudas of the Pain Unit collaborated with Dr. Azucena García Palacios and Dr. Diana Castilla López of the Universitat Jaume I in the final development of the application of pain, Following the guidelines of Rosser and Eccleston. App content validity and usability was tested in a previous study at the pain unit of the Vall d'Hebron Hospital (Suso-Ribera et al., in preparation). Thus, the study objective is to test if the introduction of this tool in the day-to-day work of the pain unit improves pain management of chronic pain patients. To do this, it is necessary to compare the evolution of patients who follow the usual treatment at the pain unit (without app) with a group of patients who do use the Pain Monitor app.

ELIGIBILITY:
Inclusion Criteria:

* The patient is over 18 years of age
* The patient has a mobile phone with Android operating system
* The patient has the physical ability to use the application
* The patient does not present psychological and / or cognitive alterations or problems with language that make their participation difficult
* The patient voluntarily wants to participate and signs the informed consent

Exclusion Criteria:

* The patient is under 18 years
* The patient does not have a mobile phone or has a mobile phone in which Android is not the operating system (the app is currently only available for Android for economic reasons)
* The patient does not have the physical capacity to use the application
* The patient does not have the capacity to participate due to psychological and / or cognitive alterations or problems with language
* The patient does not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity by an 11-point Numerical Rating Scale | First study day and end of study (Day 1 and day 30)
  Level of pain intensity experienced by the patient. Measure: Brief pain intensity questionnaire. 0-10 range (0=no pain, 10=maximum pain)
Change in side effects | First study day and end of study (Day 1 and day 30)
  A list of the most frequent side effects of pain medication has been created. Dicotomous variable. For each side effect: 0=side effect not present; 1=side effect present

SECONDARY OUTCOMES:
Change in pain interference by an 11-point Numerical Rating Scale | First study day and end of study (Day 1 and day 30)
  Interference of pain with patient's life. Brief Pain Inventory questionnaire. 0-10 range (0=no interference, 10=maximum interference)
Change in depression | First study day and end of study (Day 1 and day 30)
  Hospital Anxiety and Depression Scale. Item scoring is 0 to 3. Response anchors vary across items. Subscale range is 0-21. Higher scores indicate more depression
Change in anxiety | First study day and end of study (Day 1 and day 30)
  Hospital Anxiety and Depression Scale. Item scoring is 0 to 3. Response anchors vary across items. Subscale range is 0-21. Higher scores indicate more anxiety
Change in pain catastrophizing | First study day and end of study (Day 1 and day 30)
  Pain Catastrophizing Scale. Item scoring is 0=not at all to 4=all the time. Scale range is 0 to 52. Higher scores indicate more catastrophizing

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario de Castelló, Castellon, Spain

REFERENCES:
- [Derived] Jaen I, Suso-Ribera C, Castilla D, Zaragoza I, Garcia-Palacios A, Gomez Palones JL. Improving chronic pain management with eHealth and mHealth: study protocol for a randomised controlled trial. BMJ Open. 2019 Dec 29;9(12):e033586. doi: 10.1136/bmjopen-2019-033586. PMID 31888939